CLINICAL TRIAL: NCT06524908
Title: Study of the Effectiveness of an Exercise Intervention Oriented Toward Fat Loss in Adolescents
Brief Title: Study on the Effectiveness of a School-Based Fat Loss Program for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aiyoudong Children and Youth Sports Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Basic-2334
Record Dates: First submitted 2024-06-27; First posted 2024-07-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-07

CONDITIONS: Prevention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and dietary calorie restriction intervention group (Experimental): Received a twelve-week comprehensive intervention. The number of participants is 50.
  Interventions: Behavioral: Exercise and dietary calorie restriction
- control group (No Intervention): Normal school life without any intervention. The number of participants is 50.

INTERVENTIONS:
Behavioral: Exercise and dietary calorie restriction — The intervention group received an exercise intervention three times a week (resistance exercise from 4:30-5:00 p.m. and aerobic exercise from 5:00-5:30 p.m.), and a caloric restriction intervention (guided semi-libre diet with caloric intake restricted to 75% of overall consumption, with parents keeping track of calories and food groups and receiving regular check-ups)
  Arms: Exercise and dietary calorie restriction intervention group

SUMMARY:
The students were divided into an intervention group and a control group. The intervention group attended fat loss exercise classes three times a week and the parents cooperated with us in dietary monitoring and control. Before and after the intervention, questionnaires were completed, physical fitness and body composition were measured, and physical activity measurement bracelets were worn for 4 days. In this study, it is possible to know the mental health state, physical activity habits, body composition and physical fitness of adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Passed PAR-Q questionnaire screening
* No professional sports experience
* Able to understand the test
* Voluntarily participate in the entire testing process

Exclusion Criteria:

* Serious organic pathology of the heart, brain, lungs, kidneys, and locomotor system
* Taking medication for a chronic condition
* Have history of psychiatric disorders
* Inability to complete follow-up visits or poor adherence.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Body fat percentage (%) | From enrollment to the end of intervention at 12 weeks
  Measured by Inbody, a body composition tester using bioelectrical impedance, in %.
Physical fitness | From enrollment to the end of intervention at 12 weeks
  Measured using China National Standards for Students' Physical Health (2014 revision), with a minimum value of 0 and a maximum value of 100, higher scores respond to better fitness.
Physical activity | From enrollment to the end of intervention at 12 weeks
  Physical activity (PA) was measured using Actigraph GT3X+ accelerometers, with data expressed as minutes per day (min/day).
Fat-free mass | From enrollment to the end of intervention at 12 weeks
  Measured by Inbody, a body composition tester using bioelectrical impedance, in kg.
Fat mass | From enrollment to the end of intervention at 12 weeks
  Measured by Inbody, a body composition tester using bioelectrical impedance, in kg.

SECONDARY OUTCOMES:
Salivary testosterone | From enrollment to the end of intervention at 12 weeks
  Salivary testosterone levels were measured using radioimmunoassay (RIA) and expressed in picograms per liter (pg/L).
Resilience | From enrollment to the end of intervention at 12 weeks
  Connor-Davidson Resilience Scale-10 (CD-RISC-10). The scale consists of 10 items, each of which has a score range of 0-4, and the total score range of the scale is 0-40, with higher scores representing greater resilience.
Self-esteem | From enrollment to the end of intervention at 12 weeks
  The Rosenberg Self-Esteem Scale was used, with a total of 10 items. Scores on the scale range from 10 to 40, with higher scores indicating higher levels of self-esteem and better outcomes.
Aggression | From enrollment to the end of intervention at 12 weeks
  Assessed using the Buss-Perry Aggression Questionnaire with a total score range of 29-145. The higher the score, the more aggressive the individual is in that area and the worse the outcome.
Eating Self-efficacy | From enrollment to the end of intervention at 12 weeks
  Eating Self-Efficacy Scale .
  The minimum score is 10 and the maximum score is 100. Higher scores indicate greater self-efficacy in eating and better outcomes.
Exercise Self-Efficacy | From enrollment to the end of intervention at 12 weeks
  Exercise Self-Efficacy Scale . The minimum score is 18 and the maximum score is 180. The higher the score, the stronger the self-efficacy in exercise and the better the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Aiyoudong Children and Youth Sports Health Research Institute, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Pan X, Liu B, Gao Y, Jiang L, Chen X, Zhao D, Wang Y, Hu H, Zhao X, Lu J, Suzuki K, Zhang Y. Causal insights into the school-family-research integrated health promotion program for overweight and obesity: the independent role of moderate-to-vigorous physical activity in body fat reduction, undermined by psychological factors. Front Nutr. 2025 Jul 29;12:1577319. doi: 10.3389/fnut.2025.1577319. eCollection 2025. PMID 40799526

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT06524908/Prot_SAP_ICF_000.pdf